CLINICAL TRIAL: NCT03731091
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multiple-Site Study to Evaluate the Therapeutic Equivalence of a Generic Calcipotriene and Betamethasone Dipropionate Topical Foam, 0.005%/0.064% (Glenmark Pharmaceuticals Ltd) to the Marketed Product Enstilar® Foam (LEO Pharma Inc.) in the Treatment of Psoriasis Vulgaris (Plaque Psoriasis)
Brief Title: To Study Generic Calcipotriene and Betamethasone Dipropionate Topical Foam, 0.005%/0.064%, in the Treatment of Psoriasis Vulgaris (Plaque Psoriasis).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Glenmark Pharmaceuticals Ltd. India (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLK-1801
Record Dates: First submitted 2018-10-31; First posted 2018-11-06 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — calcipotriene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Calcipotriene/ betamethasone dipropionate topical foam (Experimental): Topical foam once daily for 4 weeks (28 days)
  Interventions: Drug: Calcipotriene/ betamethasone dipropionate topical foam, 0.005%/0.064%
- Enstilar® (Active Comparator): Topical foam once daily for 4 weeks (28 days)
  Interventions: Drug: Enstilar® foam (LEO Pharma Inc.)
- Placebo (Placebo Comparator): Topical foam once daily for 4 weeks (28 days)
  Interventions: Other: Placebo of Calcipotriene/ betamethasone dipropionate topical foam

INTERVENTIONS:
Drug: Calcipotriene/ betamethasone dipropionate topical foam, 0.005%/0.064% — Once daily for 4 weeks (28 days)
  Arms: Calcipotriene/ betamethasone dipropionate topical foam
Drug: Enstilar® foam (LEO Pharma Inc.) — Once daily for 4 weeks (28 days)
  Arms: Enstilar®
Other: Placebo of Calcipotriene/ betamethasone dipropionate topical foam — Once daily for 4 weeks (28 days)
  Arms: Placebo

SUMMARY:
A Phase III, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multiple-Site Study to Evaluate the Therapeutic Equivalence of a Generic Calcipotriene and Betamethasone Dipropionate Topical Foam, 0.005%/0.064% (Glenmark Pharmaceuticals Ltd) to the Marketed Product Enstilar® Foam (LEO Pharma Inc.) in the Treatment of Psoriasis Vulgaris (Plaque Psoriasis)

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant, non-lactating female subjects aged at least 18 years at Visit 1.
2. A clinical diagnosis of stable (at least 6 months) psoriasis vulgaris involving 5% to 30% body surface area (BSA), not including the face, axilla and groin.
3. A PGA of disease severity of at least moderate disease severity (Grade ≥ 3).
4. A plaque elevation of at least moderate severity (Grade ≥ 3) at the target lesion site. The most severe lesion at baseline should be identified as the target lesion.
5. Provide written informed consent. -

Exclusion Criteria:

1. Current diagnosis of unstable forms of psoriasis in the treatment area including guttate, erythrodermic, exfoliative, or pustular psoriasis.
2. Other inflammatory skin disease in the treatment area that may confound the evaluation of the psoriasis vulgaris (e.g., atopic dermatitis, contact dermatitis, tinea corporis).
3. Presence of pigmentation, extensive scarring, pigmented lesions, or sunburn in the treatment areas that could interfere with the rating of efficacy parameters.
4. History of psoriasis unresponsive to topical treatments.
5. History of hypersensitivity to any component of the Test or Reference product.
6. Current or past history of hypercalcemia, calcium metabolism disorder, vitamin D toxicity, severe renal insufficiency, or severe hepatic disorders.
7. Current immunosuppression.
8. Use within 6 months prior to baseline of biologic treatment for psoriasis (e.g., infliximab, adalimumab, alefacept).
9. Use within 3 months prior to baseline of: 1) chemotherapy or 2) radiation therapy.
10. Use within 2 months prior to baseline of: 1) immunosuppressive drugs (e.g., tacrolimus, pimecrolimus) or 2) oral retinoids.
11. Use within 1 month prior to baseline of: 1) systemic steroids, 2) systemic antibiotics, 3) other systemic antipsoriatic treatment, 4) psoralen and ultraviolet A (PUVA) therapy, 5) ultraviolet B (UVB) therapy, or 6) systemic anti-inflammatory agents. Note: a) Non-steroidal anti-inflammatory drugs (NSAIDs) and aspirin use on an as-needed basis and if not used consecutively for > 14 days prior to baseline and/or during the study is acceptable. Low-dose (81 mg) aspirin taken daily is acceptable. b) Intranasal or inhaled corticosteroids are acceptable if kept constant throughout the study. Intra-articular steroid injections are permissible.
12. Use within 2 weeks prior to baseline of: 1) topical antipsoriatic drugs (e.g., salicylic acid, anthralin, coal tar, calcipotriene, tazarotene), 2) topical corticosteroids, or 3) topical retinoids.
13. Use within 2 weeks prior to baseline of: 1) vitamin D supplements 2) vitamin D analogs at a dose >400 IU/day; or 3) calcium supplements (including multivitamins containing calcium).
14. Started beta-blocker therapy, antimalarial products, and/or lithium within 3 months of baseline. Subjects who have been on a steady dose for at least 3 months prior to baseline and will remain on the same dose throughout the study are eligible for study participation.
15. Subjects with planned phototherapy and/or exposure to ultraviolet A (UVA) and/or UVB during the study.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 494 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects in each treatment group with treatment success | Day 29
  Treatment success defined as none or minimal disease , a score of 0 or 1, within the treatment area(s) on the PGA scale of disease severity
The proportion of subjects in each treatment group with clinical success | Day 29
  Clinical success defined as clear or almost clear, a score of 0 or 1, at the target lesion site on the PASI scale. Each psoriatic sign of scaling, erythema, and plaque elevation should have a score of 0 or 1

CONTACTS AND LOCATIONS:
Overall Officials: William Todd Kays, Study Director — Glenmark Pharmaceuticals
Locations (30):
- United States (30):
  - Investigational Site 20, Encinitas, California
  - Investigational Site 18, Fountain Valley, California
  - Investigational Site 19, San Diego, California
  - Investigational Site 15, San Diego, California
  - Investigational Site 23, San Diego, California
  - Investigational Site 17, Santa Ana, California
  - Investigational Site 22, Santa Monica, California
  - Investigational Site 29, Clearwater, Florida
  - Investigational Site 27, Coral Gables, Florida
  - Investigational Site 1, Miami, Florida
  - Investigational Site 26, Pinellas Park, Florida
  - Investigational Site 10, New Albany, Indiana
  - Investigational Site 3, Overland Park, Kansas
  - Investigational Site 16, Louisville, Kentucky
  - Investigational Site 21, Saint Joseph, Missouri
  - Investigational Site 12, Henderson, Nevada
  - Investigational Site 28, New York, New York
  - Investigational Site 4, High Point, North Carolina
  - Investigational Site 24, Wilmington, North Carolina
  - Investigational Site 8, Beachwood, Ohio
  - Investigational Site 2, Cincinnati, Ohio
  - Investigational Site 13, Greenville, South Carolina
  - Investigational Site 7, Knoxville, Tennessee
  - Investigational site 31, Murfreesboro, Tennessee
  - Investigational Site 25, Nashville, Tennessee
  - Investigational Site 5, Austin, Texas
  - Investigational Site 11, San Antonio, Texas
  - Investigational Site 14, San Antonio, Texas
  - Investigational Site 30, Webster, Texas
  - Investigational Site 6, Norfolk, Virginia